CLINICAL TRIAL: NCT07020000
Title: A Multi-Center Post-Marketing Data Collection Protocol to Evaluate the Safety, Performance, and Health Economics of the Endoscopic Assisted Retropsoas (EARP) Interbody System for Lumbar Interbody Fusion Surgery
Brief Title: The Objective of the Protocol is to Generate Real World Evidence (RWE) Supporting the Safety, Performance, and Health Economics of Using the Regulatory Approved and Commercially Available EARP Interbody System Used During Lumbar Interbody Fusion (LIF) Procedures With the EARP Nerve Cuff Electrode
Acronym: EARP-2
Status: Not yet recruiting | Type: Observational
Sponsor: Retropsoas Technologies, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: EARP-2-1002
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Transforaminal Lumbar Interbody Fusion Surgery
Keywords: Transforaminal Lumbar Interbody Fusion Surgery; TLIF; EARP; Retropsoas Technologies, LLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Device: Nerve Cuff and Retractor System — Endoscopic Assisted Retropsoas (EARP) Nerve Cuff Electrode and an EARP Retractor system to safely monitor lumbar nerve root activity and function during standard interbody fusion surgeries.

SUMMARY:
The goal of the trial is to generate data to support the safety, performance, and cost effectiveness of using the EARP devices during Lumbar Interbody Fusion (LIF) procedures.

The primary objectives are:

* To evaluate the safety of the EARP surgical technique and devices during LIF surgeries.
* To understand the EARP fusion system's ability to achieve fusion and improve disk space over time.

DETAILED DESCRIPTION:
This multi-center post-marketing study will include consecutive patients who meet eligibility criteria, are scheduled to undergo a LIF procedure using the EARP Interbody System and EARP Nerve Cuff Electrode, and agree to participate. The study will include patients deemed appropriate for the procedure per the site's judgment, which may include patients with off-label use of the devices. Patients who consent to study participation and meet study criteria will undergo surgery according to site standard procedure. The EARP Nerve Cuff Electrode will be used to monitor nerve roots during surgery. Radiographic imaging will document the fusion status and various disk space parameters, and the Oswestry Disability Index (ODI) will be used to assess function and pain. Data will be collected from standard site follow-up visits at 6 weeks, 3 months, 6 months, and 12 months after surgery. Economic data will be collected to quantify the economics of the EARP Interbody System for LIF procedures.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing LIF between L2-S1

Exclusion Criteria:

* BMI >40 kg/m2
* Pregnant or plans on becoming pregnant in the near future
* Surgery requires combination of EARP with another lumbar interbody fusion technique (PLIF, TLIF, ALIF, OLIF, LLIF) or posterolateral fusion at another level
* History of lumbar interbody pseudoarthrosis at planned operative level
* Lumbar spondylolisthesis ≥ grade 3
* Osteoporotic vertebral compression fracture treated or untreated at planned operative site
* History of lumbar spinal metastasis
* Acute lumbar spine trauma requiring immediate intervention
* Owestry Disability Index (ODI) 81-100%
* Presence of personality disorder or major psychiatric illness
* History of allergy to titanium, platinum, PEEK, aluminum, stainless steel or silicone
* Any additional factor that makes the patient an unsuitable candidate for the study in the opinion of the principal investigator

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing LIF between L2-S1and surgeon feels is a good candidate for the EARP Procedure
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic measurements prior to surgery and at follow-up visits | From enrollment until the end of follow-up at 12 months
  Radiographic measurements including X-Ray, CT Scans, and MRIs if available
To evaluate the safety of the EARP surgical technique and devices used during LIF surgeries | From surgery until the end of follow up at 12 months
  Adverse Device Events and surgical complications due to the devices

SECONDARY OUTCOMES:
Assess the ability of the EARP fusion system to reduce pain and restore function | Baseline to final follow-up visit at 12 months
  The Oswestry Disability Index (ODI)
Assess IONM data during procedure related to the effectiveness of the EARP Nerve Cuff Electrode | During Surgery
  IONM data during surgical procedure
Quantify health economic factors associated with the EARP fusion system for LIF procedures | From surgery to end of follow up at 12 months
  Health economic data including OR time, operative time, hospital length of stay, anesthetic technique, unilateral vs. bilateral fixation, bone graft choice

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwell/Phelps, Sleepy Hollow, New York
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - Alleghany Health Network, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  For individual participant data meta-analysis.
  Information can be accessed by contacting the Sponsor directly (contact info TBD)
URL: https://www.inquiry-research.com/